CLINICAL TRIAL: NCT03577379
Title: Vascular Changes of Rotator Cuff Repair Augmented With a Whole Blood Fibrin Clot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Barbara Cottage Hospital (Other)
Responsible Party: Principal Investigator, Christopher Proctor, Managing Partner, Alta Orthopaedics, Santa Barbara Cottage Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 17-34
Record Dates: First submitted 2018-06-23; First posted 2018-07-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff repair, whole blood fibrin clot
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will be randomized to either the treatment or control group using an automated randomization program using a research electronic data capture (REDCap) system prior to surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the control arm will receive standard of care for their rotator cuff tear, and will not receive the additional whole blood fibrin clot.
- Treatment (Experimental): Patients in the control arm will receive standard of care for their rotator cuff tear, in addition to, the whole blood fibrin clot.
  Interventions: Other: Whole Blood Fibrin Clot

INTERVENTIONS:
Other: Whole Blood Fibrin Clot — For all patients assigned to the treatment group, 35mL of whole blood will be obtained during surgery by an anesthesiologist. 5 mL of the blood will be sent for pre-clot formation cell count evaluation for platelets, red blood cells and white blood cells. The remaining 30mL will be placed into a sterile container with a sintered glass cylinder supported by the lid for fibrin clot formation. The clot formation cups will be placed on a rotator at room temperature for 10 minutes at 125rpm. The fibrin clot will be removed and 5mL of the post-clot serum sent for post-clot formation cell count evaluation for platelets, red blood cells, and white blood cells.
  Arms: Treatment

SUMMARY:
The goal of this study is to assess whether undergoing surgical repair of the rotator cuff with the additional intervention of whole blood fibrin clot will improve rotator cuff vascularization at the bone-tendon interface repair site and patient outcomes compared to those who do not receive the whole blood fibrin clot intervention.

DETAILED DESCRIPTION:
Patient outcomes after rotator cuff repair vary greatly and depend on the size of the tear itself. Researchers have identified a number of devices that can be used to reinforce the surgical repair and enhance the structure and function of both the muscles and tendons (Jo et al., 2011; Randelli, Arrigoni, Ragone, MEng, Aliprandi, Cabitza, 2011; Proctor, 2014). Reinforcement patches have been used to help improve surgical outcomes, including: allograft rotator cuff, human cadaveric skin, pig and bovine skin, equine pericardium, and porcine intestinal submucosa (Randelli, Arrigoni, Ragone, MEng, Aliprandi, Cabitza, 2011). Although synthetic patches have also shown some effectiveness, these patches do not provide biologic augmentation of the tendon repair (Jo et al., 2011).

Additionally, there has been some research examining the effectiveness of using platelet-rich plasma therapy to help repair both rotator cuff tendinopathy and tears. Platelets play an important role in the healing process and it has been theorized that exposing inflamed or healing tissue to higher densities of platelets can contribute to less pain, better range of motion (ROM), and overall healing (Pandey et al., 2016). The consensus on this type of therapy has shown inconclusive results, however. For example, research by Jo et al. (2011) found no significant change in clinical recovery in respect to pain or ROM compared to a control group. Alternatively, Pandey et al. (2016) found significant improvements in both pain and ROM scores as well as decreased re-tear rates in the plasma-rich protein treatment group. These and other similar studies utilized different methodologies for patient populations (tendinopathy versus full tears, etc.), treatment timing, formulation of platelet-rich plasma or whole blood fibrin clot, and time of follow-up. Further research is needed to identify what treatments, if any, in the field of platelet-rich plasma are most beneficial for patients with rotator cuff tears. Recent research has demonstrated that whole blood fibrin clots concentrate 98% of available platelets and release growth factors including vascular endothelial growth factor over two weeks (Siegel, Clevenger, Proctor, Clegg, & Proctor, 2017). However, clinical evidence indicating the effect of whole blood fibrin clots on the healing of repaired torn rotator cuffs is lacking (Jo et al., 2011). The goal of this study is to assess whether undergoing surgical repair of the rotator cuff with the additional intervention of whole blood fibrin clot will improve rotator cuff vascularization at the bone-tendon interface repair site and patient outcomes compared to those who do not receive the whole blood fibrin clot intervention.

ELIGIBILITY:
Inclusion Criteria:

1) Presence of ultrasonographic or magnetic resonance imaging (MRI) documented rotator cuff tear confirmed at surgery to be a medium to large-sized rotator cuff tear (> 1 cm), which requires intervention due to persistent difficulty in elevation of affected shoulder and/or pain; 2) ability to give informed consent for procedure, rehabilitation, and regular clinical and radiologic follow-up for a minimum period of 6 most post-surgery; and have 3) preoperative blood platelet counts >150,000/microliter.

Exclusion Criteria:

1) they have a type III subscapularis tear and above due to different rehabilitation protocol; 2) massive, partial, or traumatic cuff tears; 3) partial or incomplete repairs; 4) is a chronic smoker or patient with Parkinson's disease; 5) have a condition that may hinder healing or attending follow-up visits (e.g., diabetes, immunocompromised status, chemotherapy treatment, chronic steroid use); and 6) age >70.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Vascularity Index | Assessed 6 weeks postoperatively.
  Vascularity or the structural outcome will be assessed at 6 weeks postoperatively using the vascularity index scoring system described in Zumstein et al., (2014).

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Assessed at baseline and at 1 week, 3 weeks, and then at 3 and 6 months.
  A 10-point pain scale for pain at night, with 0 being no pain and 10 being unbearable.
Western Ontario Rotator Cuff Index | Assessed at baseline, and 3 and 6 months.
  A 21 - item questionnaire that measures quality of life for patients with rotator cuff disease.
Veterans Rand (VR-12) | Assessed at baseline, and 3 and 6 months.
  A generic quality of life measure that consists of 12 items.
American Shoulder and Elbow Surgeons Score (ASES) | Assessed at baseline and at 3 and 6 month.
  A 100-point scale which measures pain (up to 50 points) and function (up to 50 points). A higher score indicates less pain and better function.
Single Assessment Numeric Evaluation Score (SANE) | Assessed at 3 and 6 months.
  A single -item questionnaire that asks "What percentage of normal is your shoulder?" A rating scale from 0% to 100% is given with higher being better.

CONTACTS AND LOCATIONS:
Locations (1):
- De La Vina Surgery Center, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No
Results on the aggregate of the sample will be published.

REFERENCES:
- [Background] Proctor CS. Long-term successful arthroscopic repair of large and massive rotator cuff tears with a functional and degradable reinforcement device. J Shoulder Elbow Surg. 2014 Oct;23(10):1508-13. doi: 10.1016/j.jse.2014.01.010. Epub 2014 Apr 13. PMID 24725892
- [Result] Proctor CS. Rotator cuff repair augmented with endogenous fibrin clot. Arthrosc Tech. 2012 May 18;1(1):e79-82. doi: 10.1016/j.eats.2012.03.002. Print 2012 Sep. PMID 23766981